CLINICAL TRIAL: NCT02383433
Title: A Phase II Study of Second-Line Therapy With Regorafenib Plus Gemcitabine in Metastatic Pancreatic Cancer
Brief Title: Regorafenib Plus Gemcitabine in Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI discretion based on low accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5214; NCI-2015-00146 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE5214 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
MeSH Terms: interventions — regorafenib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (regorafenib, gemcitabine hydrochloride) (Experimental): Patients receive regorafenib PO QD on days 1-21 and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Regorafenib; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Regorafenib — Given PO
  Other Names: BAY 73-4506; multikinase inhibitor BAY 73-4506; Stivarga
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdC; dFdCyd

SUMMARY:
This phase II trial studies how well regorafenib and gemcitabine hydrochloride work as second-line therapy (treatment given when initial treatment doesn't work) in treating patients with pancreatic cancer that has spread to other parts of the body. Regorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving regorafenib together with gemcitabine hydrochloride may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy (progression-free survival) of regorafenib and gemcitabine (gemcitabine hydrochloride) in previously treated patients with metastatic pancreatic cancer.

SECONDARY OBJECTIVES:

I. To assess the safety of regorafenib in combination with gemcitabine. II. To assess response rate (RR). III. To assess overall survival (OS).

OUTLINE:

Patients receive regorafenib orally (PO) once daily (QD) on days 1-21 and gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up to 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic pancreatic adenocarcinoma (or any mixed pathology if adenocarcinoma is predominant)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan
* Prior Therapies: Patients must have received at least one prior systemic chemotherapy regimen for metastatic pancreatic cancer. They should have experienced disease progression or intolerable toxicity from that regimen.
* Patients who have received prior non-gemcitabine-based systemic chemotherapy for metastatic disease at any time 4 weeks prior to enrollment, or those who are beyond 12 months of exposure to gemcitabine-based chemotherapy regimen are allowed.
* Prior chemotherapy, radiation therapy, concurrent chemoradiation are allowed if used for treatment of non-metastatic disease.
* Any chemotherapy must have been completed 4 weeks prior to enrollment
* Any radiotherapy must have been completed 2 weeks prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy of at least 12 weeks (3 months)
* Subjects must be able to understand and be willing to sign the written informed consent form; a signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure
* All acute toxic effects of any prior treatment have resolved to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version (v)4.0 grade 1 or less at the time of signing the informed consent form (ICF)
* Total bilirubin =< 1.5 x the upper limits of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Alkaline phosphatase limit =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Lipase =< 1.5 x the ULN
* Serum creatinine =< 1.5 x the ULN
* International normalized ratio (INR)/partial thromboplastin time (PTT) 1.5 x ULN; (subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in coagulation parameters exists; close monitoring of at least weekly evaluations will be performed until INR/PTT is stable based on a measurement that is pre-dose as defined by the local standard of care)
* Platelet count >= 100000/mm^3, hemoglobin (Hb) ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1500/mm^3; blood transfusion to meet the inclusion criteria will not be allowed
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug; post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 3 months after the last dose of study drug; the definition of adequate contraception will be based on the judgment of the principal investigator or a designated associate
* Subject must be able to swallow and retain oral medication

Exclusion Criteria:

* Chemotherapy within 4 weeks prior to entering the study, radiotherapy within 2 weeks prior to entering the study or failure to recover from adverse events to grade 1 or less due to agents administered more than 4 weeks earlier
* Use of any other investigational agents
* Previous assignment to treatment during this study; subjects permanently withdrawn from study participation will not be allowed to re-enter study
* Uncontrolled hypertension (systolic pressure > 140 mm Hg or diastolic pressure > 90 mm Hg [NCI-CTCAE v4.0] on repeated measurement) despite optimal medical management
* Active or clinically significant cardiac disease including:

  * Congestive heart failure - New York Heart Association (NYHA) > class II
  * Active coronary artery disease
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
  * Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization
* Evidence or history of bleeding diathesis or coagulopathy
* Any hemorrhage or bleeding event >= NCI CTCAE grade 3 within 4 weeks prior to start of study medication
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of informed consent
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology from pancreatic cancer except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor; subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed; all cancer treatments must be completed at least 3 years prior to study entry (i.e., signature date of the informed consent form)
* Patients with phaeochromocytoma
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy
* Any infection requiring ongoing intravenous antibiotics for management
* Symptomatic metastatic brain or meningeal tumors; treated and stable, asymptomatic brain metastases, as long as treatment was greater than 4 weeks prior to informed consent, are allowed
* Presence of a non-healing wound, non-healing ulcer, or bone fracture
* Renal failure requiring hemo-or peritoneal dialysis
* Dehydration grade >= 1 NCI-CTCAE v4.0
* Patients with seizure disorder requiring medication
* Persistent proteinuria >= grade 3 NCI-CTCAE v4.0 (> 3.5 g/24 hrs, measured by urine protein:creatinine ratio on a random urine sample)
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent
* Pleural effusion or ascites that causes respiratory compromise (>= NCI-CTCAE version 4.0 grade 2 dyspnea)
* History of organ allograft (including corneal transplant)
* Known or suspected allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial
* Any malabsorption condition
* Women who are pregnant or breast-feeding
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davendra Sohal, MD, MPH, Principal Investigator — Case Comprehensive Cancer Center; Jennifer Eads, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Regorafenib, Gemcitabine Hydrochloride)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Disease progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Regorafenib, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time-to-event data will be summarized using the Kaplan-Meier method.
Time Frame: Up to 1 year from enrollment
Population: Data was not collected for this outcome, study terminated early due to low accrual.
Arm/Group | Treatment (Regorafenib, Gemcitabine Hydrochloride)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected up to 3 months while on treatment.
Arm/Group | Treatment (Regorafenib, Gemcitabine Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Regorafenib, Gemcitabine Hydrochloride) (N=2)
Neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Hepatic Vein Thrombus (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Regorafenib, Gemcitabine Hydrochloride) (N=2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
alkaline phosphatase, increased gr1 (Investigations) | 1 (1)
ALT increased (Investigations) | 1 (8)
ALT increased, gr1 (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
AST increased (Investigations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
decreased platelets (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hepatic Vein Thrombosis (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia, gr1 (Metabolism and nutrition disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
increased ALT (Investigations) | 1 (1)
Increased creatinine (Investigations) | 1 (1)
Increased Lipase (Investigations) | 1 (1)
Infections, other : Thrush mouth (Infections and infestations) | 1 (1)
Intermittent Fatigue (General disorders) | 1 (1)
Intermittent Hypertension (Vascular disorders) | 1 (1)
Intermittent Nausea (Gastrointestinal disorders) | 1 (1)
Leukopenia, gr1 (Investigations) | 1 (1)
Lymphocyte Count decreased (Investigations) | 1 (1)
muscle soreness, R shoulder, gr1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
neutropenia (Investigations) | 1 (1)
Petechial Rash, gr1 (Skin and subcutaneous tissue disorders) | 1 (1)
platelet count decreased (Investigations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (2)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
pruritis, gr1 (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus Pain (Nervous system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
sunburn (Skin and subcutaneous tissue disorders) | 1 (1)
Thombocytopenia (Investigations) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1)
Thrombocytopenia, gr1 (Investigations) | 1 (1)
Weight Gain (Investigations) | 1 (1)
Weight Loss (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
worsening hypertension, gr2 (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Data was not collected, study terminated early due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT02383433/Prot_SAP_001.pdf